CLINICAL TRIAL: NCT05480787
Title: Pharmacokinetic Study of Continuous Infusion of Remazolam in Mechanically Ventilated Patients in ICU : Establishment of Population Pharmacokinetic Model and Exploration of Clinical Influencing Factors
Brief Title: Pharmacokinetic Study of Continuous Infusion of Remazolam in Mechanically Ventilated Patients in ICU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020120989remimazolam
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Intensive Care Unit; Mechanical Ventilation; Anesthesia; Liver Failure; Pharmacokinetics
Keywords: Remimazolam; Intensive Care Unit; Mechanical Ventilation; Anesthesia; Sedation; Liver Failure; Pharmacokinetics
MeSH Terms: conditions — Liver Failure | interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam 0.1mg/kg/h (Experimental): Participants were first induced with 5mg in 1-min intravenous injection and then maintained at 0.1 mg/kg/h.
  Interventions: Drug: Remimazolam 0.1mg/kg/h
- Remimazolam 0.3mg/kg/h (Experimental): Participants were first induced with 5mg in 1-min intravenous injection and then maintained at 0.3 mg/kg/h.
  Interventions: Drug: Remimazolam 0.3mg/kg/h
- Remimazolam 0.5mg/kg/h (Experimental): Participants were first induced with 5mg in 1-min intravenous injection and then maintained at 0.5 mg/kg/h.
  Interventions: Drug: Remimazolam 0.5mg/kg/h

INTERVENTIONS:
Drug: Remimazolam 0.1mg/kg/h — Remimazolam Tosilate for Injection(36mg)
  Arms: Remimazolam 0.1mg/kg/h
Drug: Remimazolam 0.3mg/kg/h — Remimazolam Tosilate for Injection(36mg)
  Arms: Remimazolam 0.3mg/kg/h
Drug: Remimazolam 0.5mg/kg/h — Remimazolam Tosilate for Injection(36mg)
  Arms: Remimazolam 0.5mg/kg/h

SUMMARY:
To study the pharmacokinetics of continuous infusion of remazolam in ICU mechanically ventilated critically ill patients, and the characteristics of PK in patients with liver failure; to explore whether liver failure affects the metabolism of remazolam by established population pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to ICU for tracheal intubation and mechanical; Patients aged >18 years; Patients with expected mechanical ventialation time >24 hours.

Exclusion Criteria:

Patients on long-term anti-anxiety medication or sleeping pills; Patients with known or suspected hypersensitivity to remimazolam; Patients with severe central nervous system diseases; Patients who do not wish to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of Remimazolam | 24 hours
  Plasma concentration of Remimazolam

SECONDARY OUTCOMES:
Adverse reactions | 28 days
  Adverse reaction that patients experience with the medication,such as hypertension,hypotension,rapid heart rate,slow heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hu J, Zhao Y, Shao L, Zhang W, Wang H, Liu Y, Su M, Zuo X. Pharmacokinetic Properties and Therapeutic Effectiveness of Remimazolam in ICU Patients With Mechanical Ventilation: A Preliminary Study. Pharmacol Res Perspect. 2025 Jun;13(3):e70130. doi: 10.1002/prp2.70130. PMID 40517312